CLINICAL TRIAL: NCT04846803
Title: Bacterial Interference for Preventing Recurrent Urinary Tract Infection - New Ways of Treatment
Acronym: BIrUTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karin Andersen, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BIrUTI
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Urinary Tract Infections
Keywords: rUTI; E.coli; prophylactic; bladder lavage
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Intervention Model Description: Inclusion with 6 months observation (standard treatment). Randomisation in ratio 3:1 for treatment initiation at baseline.
  1. Patients with prophylactic bladder flushing with an ABU strain.
  2. The control group with saline bladder flushing .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients prophylatic treated with ABU (Experimental): Patients with prophylactic bladder flushing with an ABU strain.
  Interventions: Biological: ABU bladder lavage
- Patients control group (Placebo Comparator): The control group with bladder flushing with saline solution.
  Interventions: Biological: Saline bladder lavage

INTERVENTIONS:
Biological: ABU bladder lavage — Clinical effect of preventive treatment (prophylactic treatment) - bladder lavage with the non-pathogenic bacterial strain (ABU)
  Arms: Patients prophylatic treated with ABU
Biological: Saline bladder lavage — Clinical effect of preventive treatment (prophylactic treatment) - bladder lavage with saline
  Arms: Patients control group

SUMMARY:
Urinary tract infection (UTI) is one of the most common bacterial infections worldwide. It affects 150 million people annually. Treatment of patients with UTI entails a high consumption of antibiotics and large social and health costs. With this protocol, we want to elucidate alternative treatment methods for especially recurrent urinary tract infection. Bacteria have internal competitiveness (bacterial interference) and it is known that the non-pathogenic E.coli can outcompete the pathogenic E.coli in laboratory studies.

We intend to strengthen the clinical evidence that it can be used as patient treatment through a clinical, placebo-controlled, double-blind trial at Odense University Hospital.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is one of the most common bacterial infections worldwide. It affects 150 million people annually. Treatment of patients with UTI entails a high consumption of antibiotics and large social and health costs. With this protocol, we want to elucidate alternative treatment methods for especially recurrent urinary tract infection. Bacteria have internal competitiveness (bacterial interference) and it is known that the non-pathogenic E.coli can outcompete the pathogenic E.coli in laboratory studies.

We intend to strengthen the clinical evidence that it can be used as patient treatment through a clinical, placebo-controlled, double-blind trial at Odense University Hospital.

Claim to be investigated:

* The non-pathogenic bacterial strain (ABU) E.coli can overcome the most common pathogenic E.coli (UPEC) in humans.
* ABU can be used for preventive treatment in patients with recurrent urinary tract infections.

Clinical effect of preventive treatment (prophylactic treatment) with the non-pathogenic bacterial strain (ABU) in a selected group of patients with recurrent cystitis: A clinical, placebo-controlled, triple-blinded study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with recurrent cystitis including 2 times of rUTI within the last 6 months or 3 times in the last 12 months, where at least 2 cultures show the same bacteria.
* Normal investigation for lower urinary tract diseases (LUTD) including voiding diary, symptom scores, flexible cystoscopy, voiding diagram and test for residual urine.
* Failed previously treatments.
* Patients with native bladder with both spontaneous voiding, the need for clean intermittent catheter (CIC) or indwelling catheter.
* Patients with neurogenic and non-neurogenic bladder dysfunction.
* Patients with urostomy, kidney transplantation or another complicated genesis.
* Written consent.

Exclusion Criteria:

* Malignancy in the urinary tract, kidney-, ureteral- or bladder stones, age < 18 years, pregnancy, breastfeeding. Patients in ongoing orally antibiotic treatment. Not able to speak or understand Danish.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of UTI events in the follow-up period | 1½ year
  The number of prescriptions or hospital visits

SECONDARY OUTCOMES:
Time to first UTI after the intervention | 1½ year
  Symptoms and the need for medical treatment or hospitalisation
Quality of life by standard Questionnaires_ICIQ-OABqol 08/04 | 1½ year
  International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life Module (ICIQ-OABqol).
  ICIQ-OABqol is a patient-completed questionnaire evaluating the quality of life (QoL) in patients with overactive bladder. It is translated into Danish and chosen because UTI symptoms often resemble OAB symptoms.
  Scoring: 25-160 overall score with greater values indicating increased impact on quality of life
O´Leary-Sant Voiding and Pain symptom score | 1½ year
  The O'Leary-Sant Interstitial Cystitis Symptom Index is translated into Danish and chosen because UTI symptoms often resemble the bladder pain symptoms. The O'Leary-Sant instrument is comprised of a Symptom Index (score range: 0-20 points) and a Problem Index (score range: 0-16 points), each of which contains four questions related to urinary and pain symptoms. For each index, the score is calculated by summing the points for each item. Overall score with greater values indicating increased symptom severity.
EQ-5D-5L | 1½ year
  Questionnaire evaluating quality of life at 5 terms (mobility, self-care, usual activities, pain, discomfort and anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. EQ-5D-5L health states may be converted into a single index value. The index values, presented in country-specific value sets, are a major feature of the EQ-5D instrument, facilitating the calculation of quality-adjusted life years (QALYs) that are used to inform economic evaluations of health care interventions.
CRF | 1½ year
  Case report form with respect to urinary/bladder symptoms, odour, perfomancestatus ect
Hospitalization | 1½ year
  Hospital visit due to UTI
Complications (bleeding, pain) | 1½ year
  Complications due to bladder lavage
Microbiological diagnostics: Etiology, resistance | 1½ year
  Measurements during treatment protocol
Creatinin | 1½ year
  Measurements during treatment protocol in micromol/L
Leukocytes and neutrofilocytes | 1½ year
  Measurements during treatment protocol in 10E9/L
Natrium and kalium | 1½ year
  Measurements during treatment protocol in mmol/L
CRP | 1½ year
  Measurements during treatment protocol in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Karin Andersen, Principal Investigator — University of Southern Denmark
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Odense University Hospital, Odense C

IPD SHARING:
Plan to Share IPD: No